CLINICAL TRIAL: NCT03573401
Title: A Randomized, Double Blind, Vehicle-controlled Multicenter Phase III Study to Evaluate the Safety and Efficacy of BF-200 ALA (Ameluz®) and BF-RhodoLED® in the Treatment of Superficial Basal Cell Carcinoma (sBCC) With Photodynamic Therapy (PDT).
Brief Title: Study to Evaluate the Safety and Efficacy of BF-200 ALA (Ameluz®) and BF-RhodoLED® in the Treatment of Superficial Basal Cell Carcinoma (sBCC) With Photodynamic Therapy (PDT).
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biofrontera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALA-BCC-CT013
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Superficial Basal Cell Carcinoma
Keywords: ALA-PDT
MeSH Terms: interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- BF-200 ALA (Experimental): Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid).
  Photodynamic therapy (PDT)
  Interventions: Combination Product: Photodynamic therapy (PDT) (ALA-PDT, Ameluz®-PDT)
- Vehicle (Placebo Comparator): Topical application of vehicle to BF-200 ALA containing no active ingredient. Photodynamic therapy (PDT)
  Interventions: Combination Product: Placebo Photodynamic therapy (PDT) (vehicle to BF-200 ALA containing no active ingredient)

INTERVENTIONS:
Combination Product: Photodynamic therapy (PDT) (ALA-PDT, Ameluz®-PDT) — The Main Target Lesion will be marked by at least 3 ink marks prior to PDT to enable precise excision for histopathological assessment 12 weeks after the first or second PDT cycle dependent on the clearance status of the lesion. All target lesions should be prepared prior to drug application by degreasing, removal of all scabs and crusts, and roughening of the surface, if appropriate. Bleeding should be avoided. The formulations will then be applied to the lesions (maximal combined lesion area incl. margin is 20 cm²) located in 1 to 2 illumination areas. The medication should be applied to the entire lesion(s) plus a 0.5 - 1.0 cm margin surrounding each lesion at a thickness of 1 mm, allowed to dry (for approximately 10 minutes), covered with occlusive dressing, and incubated for approximately 3 h. Thereafter, any remnants of the IMP will be removed carefully and the PDT illumination will be administered using the light emitting diode (LED) red light device BF-RhodoLED®.
  Other Names: ALA-PDT, Ameluz®-PDT
  Arms: BF-200 ALA
Combination Product: Placebo Photodynamic therapy (PDT) (vehicle to BF-200 ALA containing no active ingredient) — The Main Target Lesion will be marked by at least 3 ink marks prior to PDT to enable precise excision for histopathological assessment 12 weeks after the first or second PDT cycle dependent on the clearance status of the lesion. All target lesions should be prepared prior to drug application by degreasing, removal of all scabs and crusts, and roughening of the surface, if appropriate. Bleeding should be avoided. The formulations will then be applied to the lesions (maximal combined lesion area incl. margin is 20 cm²) located in 1 to 2 illumination areas. The medication should be applied to the entire lesion(s) plus a 0.5 - 1.0 cm margin surrounding each lesion at a thickness of 1 mm, allowed to dry (for approximately 10 minutes), covered with occlusive dressing, and incubated for approximately 3 h. Thereafter, any remnants of the IMP will be removed carefully and the PDT illumination will be administered using the light emitting diode (LED) red light device BF-RhodoLED®.
  Arms: Vehicle

SUMMARY:
The aim of this study is to test the safety and efficacy of photodynamic therapy (PDT) with the medication Ameluz® performed with the PDT-lamp BF-RhodoLED® in comparison to the respective placebo treatment for superficial basal cell carcinoma (BCC).

DETAILED DESCRIPTION:
The study will be conducted as randomized, double blind and vehicle-controlled ( 4:1 ratio of verum (BF-200 ALA; Ameluz®) to vehicle (placebo)) clinical trial at 15 sites in the United States of America (US). Each site should randomize between 10 and 20 subjects.

Each subject will complete a clinical observation period that will last for up to 7 months (up to 4 weeks screening and pre-randomization period, and up to 6 months clinical observation period) followed by a 5-year follow-up (FU) period after the completion of the first PDT cycle.

The treatment of superficial BCC lesion(s) comprises of up to two PDT cycles each with two PDT sessions one to two weeks apart of each other. 12 weeks after the first PDT of the first cycle lesion(s) will be assessed clinically and only subjects with remaining BCC lesion(s) will be retreated in the second PDT cycle starting the same day. For clinically completely cleared subjects the clinical observation period of the study will end and these subjects will enter the FU part of the study.

For each subject a Main Target Lesion will be defined that will be excised either 12 weeks after the first PDT of the first cycle, if clinically cleared, or at the end of the clinical observation period in order to histologically confirm the clinical assessment. Additional Target Lesions will be assessed clinically, only. Randomization will be stratified by the number of lesions (1 vs ≥2 Lesion(s)).

Definitions of complete responders comprise of:

1. Complete response of the Main Target Lesion which is assessed 12 weeks after the start of the last PDT cycle that included treatment of the Main Target Lesion and is defined as a Main Target Lesion that is completely clinically and histologically cleared.
2. In general, clinically complete responders are categorized 12 weeks after the start of the last PDT cycle according to clinical assessment only and are defined as subjects with all lesions (Main plus Additional Target Lesions) clinically cleared.

Verum and vehicle are indistinguishable. However, treatment is accompanied with typical adverse events (AEs). In order to guarantee the blind status of the investigator assessing efficacy after each PDT cycle, a second investigator or delegated person will perform drug application and light treatment as well as all safety evaluations at visits where PDT is applied and during the phone call 1 week after each PDT cycle, respectively. Both investigators (delegated person(s)) are not entitled to exchange information about the study outcome and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to sign the informed consent form and Health Insurance Portability and Accountability Act (HIPAA) form. A study-specific informed consent form and a HIPAA form must be obtained in writing for all subjects prior to starting any study procedures.
* Men or women ≥18 years of age.
* Presence of ≥1 naïve sBCC lesion in the treatment areas face/forehead, bald scalp, extremities and/or neck/trunk, all of which are, according to the clinical judgement of the investigator, likely to be histologically confirmed as sBCCs. Lesions should not be within the embryonic fusion planes (H-zone), especially within 2 cm of the hair zone or on the ears. In case of multiple lesions, one lesion is defined as Main Target Lesion which will be excised at the end of the clinical observation period. Only eligible naïve sBCCs, confirmed by histology taken at screening, are allowed to be included in the study as Main or Additional Target Lesions. Thus, eligible sBCCs must lack any histological evidence of aggressive growth patterns (e.g. severe squamous metaplasia, infiltrative/desmoplastic features or basosquamous features). BCCs assessed as non-naïve (e.g. previously treated or recurrent) or non-eligible by biopsy taken at screening (and in a distance >5 cm from the next lesion included in the study) should be excised by surgery or removed by cryotherapy in a timely manner. Other treatments for these lesions are not allowed during the study.
* The diameter of each eligible lesion should be ≥ 0.6 cm, and the entire treatment field must not exceed ~20 cm². The treatment field is defined as the field to which IMP is applied, usually including the target lesions and margins surrounding the lesions of up to 1 cm. For the Main Target Lesion, the maximal lesion size should be such that surgical excision without a skin transplant is feasible according to the investigator's judgement.
* Target BCC lesions must be discrete and located within 1-2 illumination areas (the illumination area is defined by the effective illumination area of the BF-RhodoLED® device with approximately 6 x 16 cm).
* Willingness to receive up to 4 PDTs within 3.5 months and excision of the Main Target Lesion either at Visit 5, if clinically cleared, or at the end of the clinical observation period 12 weeks after the start of the last PDT cycle (Visit 8), irrespective of whether the treated Main Target Lesion was clinically cleared or not.
* Free of significant physical abnormalities (e.g. tattoos, dermatoses) within the potential treatment field plus a 5 cm radius surrounding the target lesion(s) as they may interfere with examination or final evaluation.
* Willingness to stop the use of moisturizers and any other cosmetics within the treatment field plus a 5 cm radius surrounding the target lesion(s) 48 hours prior to an office visit and 48 hours after each PDT session. Sunscreen will be allowed, but should not be applied to the treatment field plus the 5 cm radius surrounding the target lesion(s) within approximately 24 h prior to a clinical visit.
* Acceptance to abstain from extensive sunbathing and the use of a solarium during the clinical observation period. Subjects with sunburn within treatment areas cannot be included until fully recovered.
* Healthy subjects and subjects with clinically stable medical conditions, including, but not limited to controlled hypertension, diabetes mellitus type II, hypercholesterolemia, and osteoarthritis, will be permitted to be included in the study if their medication is not prohibited by this protocol.
* Women of childbearing potential are permitted to participate in this study only if they have a negative serum pregnancy test at screening and are willing to use a highly effective method of contraception during the clinical observation period of the study.

Exclusion Criteria:

* History of hypersensitivity to 5-ALA or any ingredient of BF-200 ALA which includes soybean phosphatidylcholine.
* Hypersensitivity to porphyrins.
* Current treatment with immunosuppression therapy.
* Presence of photodermatoses.
* Presence of porphyria.
* Presence of clinically significant inherited or acquired coagulation defect.
* Evidence of clinically significant (CS) unstable medical conditions, such as:

  * Metastatic tumor or tumor with high probability of metastasis.
  * Cardiovascular disease class III, IV (New York Heart Association [NYHA]).
  * Immunosuppressive condition.
  * Hematologic, hepatic, renal, neurologic, or endocrine condition.
  * Collagen-vascular condition.
  * Gastrointestinal condition.
* Clinically relevant cardiovascular, hepatic, renal, neurologic, endocrine, or other major systemic diseases that complicate implementation of the protocol or interpretation of the study results.
* Gorlin Syndrome or Xeroderma pigmentosum.
* Presence and/or physical treatment of skin tumors other than (naïve) sBCC (e.g. malignant melanoma, squamous cell carcinoma (SCC), Bowen's disease, aggressive BCC or nBCC diagnosed at the screening visit by clinical assessment) within a distance of ≤ 5 cm from the nearest target lesion within 4 weeks prior to PDT (Visit 2) until the end of the clinical observation period. However, biopsied lesion(s) that were not confirmed eligible at screening and which are located at a distance of > 5 cm from any lesion(s) that will be included in the study can be surgically removed. Treatment by PDT or topical medication during the course of the clinical observation period of the study triggers exclusion of the subject.
* If lesion(s) are assessed as non-eligible by biopsy during initial screening and these lesions are localized within a distance of 5 cm from an otherwise suitable lesion, this suitable lesion must be excluded from the study.
* Αny AK lesions within the treatment field (lesion area including margin of 0.5 to 1.0 cm).
* Any topical medical treatment of AK, other non-melanoma skin cancers (NMSC), or melanoma (except for IMP treatment of the target lesion(s)) starting 12 weeks prior to Visit 2 (PDT-1) and lasting until the end of the clinical observation period.
* Any other topical medical treatment of the skin 12 weeks prior to Visit 2 (PDT-1) until the end of the clinical observation period, with the exception of:

  * Topical treatments with corticosteroids (allowed throughout the clinical observation period of the study).
  * Topical non-steroidal anti-inflammatory drugs (NSAIDs such as diclofenac) (allowed throughout the clinical observation period of the study with the restriction of 7 days prior to and 7 days after PDTs).
* Start of intake of medication with hypericin or systemically acting drugs with phototoxic or photoallergic potential within 8 weeks prior to screening.
* Any of the systemic treatments listed below, within the designated period prior to PDT and during the clinical observation period.

  * Interferon - 6 weeks
  * Immunomodulators or immunosuppressive therapies - 12 weeks
  * Cytotoxic drugs - 6 months
  * Investigational drugs - 8 weeks
  * Drugs known to have major organ toxicity - 8 weeks
  * Corticosteroids (oral or injectable) - 6 weeks
  * MAL or ALA - 12 weeks
* Systemic treatment with NSAIDs is not to be used 7 days prior to and 7 days after PDT. ASA (e.g. Aspirin®) up to 100 mg/ day, ibuprofen up to 200 mg/ day, and acetaminophen (e.g. Tylenol®) is allowed during this period.
* Presence of tattoos, skin inflammation, wounds, etc. in the treatment field(s) plus a 5 cm radius surrounding the target lesion(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2029-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Pariser, MD, Principal Investigator — Virginia Clinical Research, Inc.
Locations (18):
- United States (18):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Alliance Dermatology & Mohs Center, Phoenix, Arizona
  - First OC Dermatology, Fountain Valley, California
  - Cosmetic Laser Dermatology, San Diego, California
  - AboutSkin Research, LLC, Greenwood Village, Colorado
  - Dermatology Associates PA of the Palm Beaches, Delray Beach, Florida
  - University of Florida Dept of Dermatology, Gainesville, Florida
  - Laser and Skin Surgery Center of Indiana, Indianapolis, Indiana
  - Henry Ford Health System, Detroit, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - The Narrows Institute for Biomedical Research and Education, Inc., Brooklyn, New York
  - Skin Search of Rochester, Inc, Rochester, New York
  - Rochester Dermatologic Surgery, Victor, New York
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Austin Institute for Clinical Research Inc., Houston, Texas
  - Austin Institute for Clinical Research Inc., Pflugerville, Texas
  - Jordan Valley Dermatology, West Jordan, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 281 subjects assessed for eligibility, 187 subjects met the inclusion criteria and were randomized to treatment.
Groups:
- BF-200 ALA: Topical Photodynamic therapy (PDT) using the red light device BF-RhodoLED® after 3h incubation of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid).
- Vehicle: Topical Photodynamic therapy (PDT) using the red light device BF-RhodoLED® after 3h incubation of vehicle to BF-200 ALA.
Period: Overall Study
Arm/Group | BF-200 ALA | Vehicle
Started | 145 | 42
Completed | 141 | 41
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Subject non-compliance with study schedule | 1 | 0
Not completed — Discontinuation of study treatment due to subject decision | 1 | 0
Not completed — Subject required prohibited medication for concomitant medical condition | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BF-200 ALA | Vehicle | Total
Number analyzed (Participants) | 145 | 42 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 15 | 96
  >=65 years | 64 | 27 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (10.8) | 66.1 (9.8) | 63.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 11 | 78
  Male | 78 | 31 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 142 | 42 | 184
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 145 | 42 | 187
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Skin type was evaluated according to Fitzpatrick criteria (Fitzpatrick 1988). Skin type is often categorized according to the Fitzpatrick skin type scale, which ranges from very fair (skin type I) to very dark (skin type VI). Genetic disposition (color of eyes, hair, etc), reaction to sun exposure and tanning habits (sun bathing, artificial tanning or tanning creams) influence the skin type.
  Participants
    I - III | 138 | 40 | 178
    IV - VI | 7 | 2 | 9
Number of target lesions [Count of Participants; unit: Participants]
  1 target lesion | 122 | 34 | 156
  more than 1 target lesion | 23 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Composite Clinical and Histological Response of the Subject's Main Target Lesion as Assessed 12 Weeks After the Start of the Last PDT Cycle That Included Treatment of the Main Target Lesion.
Description: Each subject had one Main Target Lesion. The composite clinical and histological response rate of the subjects' Main Target Lesions is the percentage of subjects with a clinically and histologically cleared Main Target lesion 12 weeks after the start of the last PDT cycle that included treatment of the Main Target Lesion (Visit 5 or Visit 8).
Time Frame: 12 weeks after the start of the last PDT cycle that included treatment of the Main Target Lesion
Population: Full analysis set
Measure: Number; unit: percentage of subjects
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
percentage of subjects | 65.5 | 4.8

2. Secondary Outcome: Main Target Lesion Clinical Response Rate (According to Clinical Assessment Only) Assessed 12 Weeks After the Start of the Last PDT Cycle
Description: 1. Key secondary endpoint: Percentage of Main Target Lesions with complete clinical clearance (i.e. according to clinical assessment only) 12 weeks after the start of the last PDT cycle.
Time Frame: 12 weeks after the start of the last PDT cycle
Population: Full analysis set
Measure: Number; unit: percentage of Main Target Lesions
Units Other Than Participants: Number of Main Target Lesions
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
Number analyzed (Number of Main Target Lesions) | 145 | 42
percentage of Main Target Lesions | 83.4 | 21.4

3. Secondary Outcome: Main Target Lesion Histological Response Rate (According to Histological Assessment Only) Assessed 12 Weeks After the Start of the Last PDT Cycle
Description: 2. Key secondary endpoint: Percentage of Main Target Lesions with complete histological clearance (i.e. according to histological assessment only) 12 weeks after the start of the last PDT cycle.
Time Frame: 12 weeks after the start of the last PDT cycle
Population: Full analysis set
Measure: Number; unit: percentage of Main Target Lesions
Units Other Than Participants: Number of Main Target Lesions
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
Number analyzed (Number of Main Target Lesions) | 145 | 42
percentage of Main Target Lesions | 75.9 | 19.0

4. Secondary Outcome: Subject Complete Clinical Response (Complete Clearance of All Target Lesions According to Clinical Assessment Only) Assessed 12 Weeks After the Start of the Last PDT Cycle.
Description: 3. Key secondary endpoint: Percentage of subjects with complete clinical clearance of all Target Lesions (i.e. according to clinical assessment only) 12 weeks after the start of the last PDT cycle.
Time Frame: 12 weeks after the start of the last PDT cycle
Population: Full analysis set
Measure: Number; unit: percentage of subjects
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
percentage of subjects | 82.1 | 21.4

5. Secondary Outcome: Subject Complete Response (Clinically and Histologically Cleared Main Target Lesion (See Above) and Complete Clinical Remission of All Additional Target Lesions) Assessed 12 Weeks After the Start of the Last PDT Cycle.
Description: 4. Key secondary endpoint: Percentage of subjects with complete clinical and histological clearance of the Main Target Lesion and complete clinical clearance of all Additional Target Lesions 12 weeks after the start of the last PDT cycle
Time Frame: 12 weeks after the start of the last PDT cycle
Population: Full analysis set
Measure: Number; unit: percentage of subjects
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
percentage of subjects | 64.1 | 4.8

6. Secondary Outcome: Lesion Complete Clinical Response Rate Per Treatment Arm (Complete Clearance of Individual Lesions (Main and Additional Target Lesions)) According to Clinical Assessment Only, Assessed 12 Weeks After the Start of the Last PDT Cycle.
Description: Further secondary endpoint: Percentage of Individual Target Lesions that are completely clinically cleared per treatment arm 12 weeks after the start of the last PDT cycle.
Time Frame: 12 weeks after the start of the last PDT cycle
Population: Full analysis set
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Number of Target Lesions
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
Number analyzed (Number of Target Lesions) | 172 | 51
percentage of target lesions | 82.6 | 21.6

7. Secondary Outcome: Main Target Lesion Complete Response (Clinically and Histologically Cleared) Assessed 12 Weeks After PDT-1.
Description: Further secondary endpoint: Percentage of Main Target Lesions that are clinically and histologically cleared 12 weeks after PDT-1.
Time Frame: 12 weeks after PDT-1
Population: Full analysis set
Measure: Number; unit: percentage of Main Target Lesions
Units Other Than Participants: Number of Main Target Lesions
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
Number analyzed (Number of Main Target Lesions) | 145 | 42
percentage of Main Target Lesions | 44.1 | 2.4

8. Secondary Outcome: Main Target Lesion Clinical Response (According to Clinical Assessment Only) Assessed 12 Weeks After PDT-1.
Description: Further secondary endpoint: Percentage of Main Target Lesions that are clinically cleared 12 weeks after PDT-1.
Time Frame: 12 weeks after PDT-1
Population: Full analysis set
Measure: Number; unit: percentage of Main Target Lesions
Units Other Than Participants: Number of Main Target Lesions
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
Number analyzed (Number of Main Target Lesions) | 145 | 42
percentage of Main Target Lesions | 57.2 | 14.3

9. Secondary Outcome: Main Target Lesion Histological Response (According to Histological Assessment Only) Assessed 12 Weeks After PDT-1.
Description: Further secondary endpoint: Percentage of Main Target Lesions that are histologically cleared 12 weeks after PDT-1.
Time Frame: 12 weeks after PDT-1
Population: Full analysis set
Measure: Number; unit: percentage of Main Target Lesions
Units Other Than Participants: Number of Main Target Lesions
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
Number analyzed (Number of Main Target Lesions) | 145 | 42
percentage of Main Target Lesions | 44.8 | 2.4

10. Secondary Outcome: Lesion Complete Clinical Response Rate Per Treatment Arm (Complete Clearance of Individual Lesions (Main and Additional Target Lesions)) According to Clinical Assessment Only, Assessed 12 Weeks After PDT-1.
Description: Further secondary endpoint: Percentage of Individual Target Lesions that are completely clinically cleared per treatment arm 12 weeks after PDT-1
Time Frame: 12 weeks after PDT-1
Population: Full analysis set
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Number of Target Lesions
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
Number analyzed (Number of Target Lesions) | 172 | 51
percentage of target lesions | 58.7 | 13.7

11. Secondary Outcome: Subject Complete Clinical Response (Complete Clearance of All Target Lesions According to Clinical Assessment Only) Assessed 12 Weeks After PDT-1.
Description: Further secondary endpoint: Percentage of subjects with complete clinical clearance 12 weeks after PDT-1.
Time Frame: 12 weeks after PDT-1
Population: Full analysis set
Measure: Number; unit: percentage of subjects
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
percentage of subjects | 54.5 | 14.3

12. Secondary Outcome: Subject Complete Response (Clinically and Histologically Cleared Main Target Lesion (See Above) and Complete Clinical Remission of All Additional Target Lesions) Assessed 12 Weeks After PDT-1..
Description: Further secondary endpoint: Percentage of subjects with complete clinical and histological clearance of the Main Target Lesion and complete clinical clearance of Additional Target Lesions 12 weeks after PDT-1.
Time Frame: 12 weeks after PDT-1
Population: Full analysis set
Measure: Number; unit: percentage of subjects
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
percentage of subjects | 41.4 | 2.4

13. Secondary Outcome: For All Target Lesions, Assessment of Esthetic Appearance by the Investigator 12 Weeks After the Start of the Last PDT Cycle, But Prior to Surgical Excision of the Main Target Lesion and Any Alternative Treatment of Additional Target Lesions.
Description: Further secondary endpoint: Investigators assessment of the esthetic appearance of all Target lesions but prior to surgical excision of the Main Target Lesion or alternative Treatment of Additional Target Lesions
Time Frame: 12 weeks after the start of the last PDT cycle
Population: Full analysis set
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Number of Target Lesions
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
Number analyzed (Number of Target Lesions) | 168 | 50
percentage of target lesions
  Very good | 61.9 | 34.0
  Good | 27.4 | 24.0
  Satisfactory | 9.5 | 28.0
  Unsatisfactory | 0.6 | 10.0
  No answer | 0.6 | 4.0

14. Secondary Outcome: Subjects' Satisfaction Regarding Esthetic Outcome and Treatment 12 Weeks After the Start of the Last PDT Cycle, But Prior to Surgical Excision of the Main Target Lesion or Alternative Treatment of Additional Target Lesions
Description: Further secondary endpoint: Subject's assessment regarding the esthetic outcome and the Treatment 12 weeeks after the start of the last PDT cycle but prior to surgical excision of the Main Target Lesion or alternative Treatment of Additional Target Lesions
Time Frame: 12 weeks after the start of the last PDT cycle
Population: Full analysis set
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Number of Target Lesions
Arm/Group | BF-200 ALA | Vehicle
Number analyzed (Participants) | 145 | 42
Number analyzed (Number of Target Lesions) | 168 | 50
percentage of target lesions
  Very good | 65.5 | 56.0
  Good | 22.6 | 18.0
  Satisfactory | 10.7 | 8.0
  Unsatisfactory | 0.6 | 10.0
  No answer | 0.6 | 8.0

ADVERSE EVENTS:
Time Frame: The collection of adverse events (AEs) started with the subjects' informed consent (≤ 4 weeks prior to the first PDT) until the end of the clinical observation period (12 weeks after start of last PDT cycle).
Description: All AEs described in the following are treatment-emergent adverse events (TEAEs). TEAEs were defined as all AEs with time of onset on or after the time of treatment with the investigational medicinal product within 4 weeks (28 days) after each PDT cycle or AEs identified to be at least possibly related to IMP or medical device. If unclear due to incomplete start time/date of AE or PDT, AEs were assumed to be TEAEs.
Arm/Group | BF-200 ALA | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/42
Serious Adverse Events (participants affected / at risk) | 3/145 | 2/42
Other Adverse Events (participants affected / at risk) | 145/145 | 35/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BF-200 ALA (N=145) | Vehicle (N=42)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BF-200 ALA (N=145) | Vehicle (N=42)
Application site discharge (General disorders) | 4 (6) | 2 (2)
Application site discolouration (General disorders) | 13 (15) | 1 (1)
Application site erosion (General disorders) | 7 (8) | 3 (6)
Application site erythema (General disorders) | 100 (228) | 16 (48)
Application site exfoliation (General disorders) | 25 (30) | 7 (13)
Application site induration (General disorders) | 25 (39) | 3 (3)
Application site oedema (General disorders) | 42 (72) | 5 (10)
Application site pain (General disorders) | 138 (785) | 12 (24)
Application site paraesthesia (General disorders) | 35 (65) | 5 (8)
Application site pruritus (General disorders) | 73 (176) | 11 (14)
Application site scab (General disorders) | 32 (42) | 2 (2)
Application site ulcer (General disorders) | 4 (4) | 1 (1)
Application site vesicles (General disorders) | 12 (12) | 1 (1)
Application site warmth (General disorders) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (16) | 4 (7)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 10 (19) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the Study and results shall not be published in any form without prior consent of Sponsor. All decisions on the timing and content of publications/ presentations will be coordinated by Sponsor. A draft of any manuscript, talks, abstracts, and all similar material shall be submitted to sponsor at least sixty (60) days before submission of the final form to any journal, scientific conference, symposium, or program review committee prior to publication or other release.

DOCUMENTS (2):
  • Study Protocol (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT03573401/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT03573401/SAP_001.pdf